CLINICAL TRIAL: NCT03691948
Title: Reducing Prescription Opioid Misuse: Dental Provider Intervention Development
Brief Title: Reducing Prescription Opioid Misuse: ROPEs Pilot Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Jenna McCauley, Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pro00082658
Record Dates: First submitted 2018-09-27; First posted 2018-10-02 (Actual); Results first posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ROPEs (Experimental)
  Interventions: Other: Responsible Opioid Prescriber Education (ROPES)
- Control (Active Comparator)
  Interventions: Other: Active Comparator Control

INTERVENTIONS:
Other: Responsible Opioid Prescriber Education (ROPES) — The ROPEs intervention is a self-guided, web-based continuing dental education intervention. Consistent with ADA recommendations, ROPEs consists of seven modules of active content: (1) Overview; (2) Background on the Opioid Epidemic; (3) Dental Pain Management and the Role of Opioids; (4) Universal Precautions Approach; (5) Screening, Monitoring, and PDMP use; (6) Providing Patient Education; and, (7) Case Vignettes. All key intervention content is delivered via video-based platform and includes downloadable practice aides and resources.
  Arms: ROPEs
Other: Active Comparator Control — An online PDF version of the Center for Disease Control Guideline for Prescribing Opioids for Chronic Pain.
  Arms: Control

SUMMARY:
This is a randomized controlled pilot trial to establish methodological feasibility and determine whether a web-based, continuing dental education intervention regarding opioid prescribing risk mitigation strategies - consistent with ADA guidelines - produces pre-to-post changes in knowledge, motivation, and behavioral skills pertaining to the use of risk mitigation strategies when prescribing opioids in dental practice. The current study involves completion of a self-report pre-test (dentists), randomization to complete ROPEs or attention control intervention, completion of a self-report post-test (immediately following intervention/control completion), and completion of 1-month self-report follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female; any race or ethnicity; age 21-85 years.
2. Able to comprehend English.
3. Be either a licensed dental practitioner currently practicing or a Resident enrolled in the College of Dental Medicine at the Medical University of South Carolina or a practicing dentist in the Charleston-county area or a licensed dental practitioner currently participating in the National Dental Practice Based Research Network (NDPBRN).
4. Report having ever prescribed an opioid analgesic to a patient
5. Must have Internet access
6. Must have a valid, usable email account
7. Must agree to complete all study measurements.

Exclusion Criteria:

1. Unable to provide informed consent due to mental or physical limitations.
2. Participation in ROPEs intervention development focus groups.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2019-12-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Jenna McCauley, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No significant pre-assignment study events occurred.
Period: Overall Study
Arm/Group | ROPEs | Control
Started | 27 | 33
Completed | 26 | 30
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Population: All participants enrolled and randomized in the study
Groups:
- Total: Total of all reporting groups
Arm/Group | ROPEs | Control | Total
Number analyzed (Participants) | 27 | 33 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.85 (10.63) | 39.91 (12.78) | 38.08 (11.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 17 | 23 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 27 | 31 | 58
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 20 | 25 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 27 | 33 | 60

OUTCOME MEASURES:

1. Primary Outcome: Methodological Feasibility: Recruitment Rate
Description: Number of participants enrolled and randomized out of the number of individuals expressing interest and receiving log-in credentials.
Time Frame: Baseline completion, approximately 2 hours
Population: 76 individuals received log-in credentials for this study.
Measure: Count of Participants; unit: Participants
Groups:
- Overall - Intervention and Control Participants: This measure of recruitment is reported for the overall study and includes participants randomized to both intervention (ROPEs) and control arms of the study.
Arm/Group | Overall - Intervention and Control Participants
Number analyzed (Participants) | 76
Participants | 60

2. Primary Outcome: Methodological Feasibility: Completion Rates
Description: Percent of Patients Completing ROPES (or control)
Time Frame: Baseline completion, approximately 2 hours
Population: All enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | ROPEs | Control
Number analyzed (Participants) | 27 | 33
Participants | 26 | 31

3. Primary Outcome: Methodological Feasibility: Follow-Up Completion Rates
Description: Percent of baseline participants completing the one-month follow-up assessment
Time Frame: Through study completion, an average of 4-6 weeks (Baseline and one-month follow-up)
Population: All enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | ROPEs | Control
Number analyzed (Participants) | 27 | 33
Participants | 26 | 30

4. Primary Outcome: Methodological Feasibility: Time to Complete Intervention
Description: Time participant takes to finish engaging with ROPES intervention or control intervention
Time Frame: Baseline completion component, approximately 90 minutes
Population: All enrolled participants who completed the intervention. Note that 1 ROPEs participant and 1 Control participant did not start/complete the intervention, thus no data was available regarding their time to completion.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | ROPEs | Control
Number analyzed (Participants) | 26 | 31
Minutes | 108 (48.02) | 21 (18.91)

5. Secondary Outcome: Change at 1-Month Follow-Up From Baseline in Knowledge Change Questionnaire Score
Description: The Knowledge Change Questionnaire was developed specifically for this study and contains five items that assess dentists' knowledge regarding: (1) dentists' role in curbing prescription opioid misuse, initiation to abuse, and diversion; (2) recent released guideline recommendations for standard pain management in dental practices; and, (3) risk mitigation strategies, such as prescription opioid misuse screening and use of their state's PDMP. One point is awarded for each correct response to items on the questionnaire. The questionnaire scale ranges from 0 (no correct items, least knowledge) to 5 (all correct items, most knowledge).
  This outcome will assess mean differences between groups in their change (from pre-test to one-month follow-up) in knowledge regarding best practices in dental opioid prescribing.
Time Frame: Through study completion, an average of 4-6 weeks (Baseline and one-month follow-up)
Population: All participants completing the pre-test and the 1-month follow-up. Note that 1 ROPEs participant was lost to follow-up and 3 Control participants were lost to follow-up.
Measure: Mean (Standard Deviation); unit: Change in score on a scale
Arm/Group | ROPEs | Control
Number analyzed (Participants) | 26 | 30
Change in score on a scale | -.19 (1.17) | .00 (1.11)
Statistical Analysis 1: Comparison: ROPEs vs Control; Test type: Superiority; p = .531, ANOVA

6. Secondary Outcome: Change at Post-test From Baseline in Knowledge Change Questionnaire Score
Description: The Knowledge Change Questionnaire was developed specifically for this study and contains five items that assess dentists' knowledge regarding: (1) dentists' role in curbing prescription opioid misuse, initiation to abuse, and diversion; (2) recent released guideline recommendations for standard pain management in dental practices; and, (3) risk mitigation strategies, such as prescription opioid misuse screening and use of their state's PDMP. One point is awarded for each correct response to items on the questionnaire. The questionnaire scale ranges from 0 (no correct items, least knowledge) to 5 (all correct items, most knowledge).
  This outcome will assess mean differences between groups in their change (from pre-test to post-test) in knowledge regarding best practices in dental opioid prescribing.
Time Frame: Single time point from pre-intervention to immediately post-intervention
Population: All participants completing the pre-test and the post-test. Note that 1 ROPEs participant was lost to follow-up and 2 Control participants were lost to follow-up.
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | ROPEs | Control
Number analyzed (Participants) | 26 | 31
change in score on a scale | 0.42 (1.10) | -0.03 (0.80)
Statistical Analysis 1: Comparison: ROPEs vs Control; Test type: Superiority; p = 0.076, ANOVA

ADVERSE EVENTS:
Time Frame: From Enrollment (completion of first item on pre-test) through 1-month post-intervention follow-up completion
Description: As this was deemed a minimal risk study by IRB of record, with the greatest risk to participants being loss of confidentiality. This study relied on non-systematic assessment, i.e., participant report of adverse or serious adverse events. No investigator initiated assessment of adverse events was conducted.
Arm/Group | ROPEs | Control
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/33
Other Adverse Events (participants affected / at risk) | 0/27 | 0/33

LIMITATIONS AND CAVEATS:
This was a pilot trial intended to demonstrate methodological feasibility. Thus, the trial was not intended to be sufficiently powered to detect significant differences between the intervention and control groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Informed Consent Form (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/48/NCT03691948/ICF_000.pdf
  • Study Protocol (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/48/NCT03691948/Prot_001.pdf
  • Statistical Analysis Plan (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/48/NCT03691948/SAP_002.pdf